CLINICAL TRIAL: NCT05388526
Title: Relationship Between Frailty and Cognitive Impairment in Patients With Parkinson's Disease or Secondary Parkinsonism.
Brief Title: Frailty and Cognitive Function in Parkinson's Disease.
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, María Cruz Sousa Fraguas, Principal Investigator. Physiotherapist., University of Oviedo
Other Study IDs: 2022-195 Parkinson´s disease.
Record Dates: First submitted 2022-05-17; First posted 2022-05-24 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Parkinsonian disorders; Frailty; Cognitive dysfunction; Cognition disorders; Home care services; Home care agencies
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Frailty; Cognitive Dysfunction; Cognition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson: Patients with a diagnosis of PD or secondary parkinsonism belonging to the Health Area V of the Health Service of the Principality of Asturias, Spain.
  Patient origin: Rehabilitation Service Instituto de Rehabilitación Astur S.A. and Asociación de Parkinson Jovellanos, from Gijón, Asturias, Spain.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention to be administered, only collection of data through various tests and questionnaires.

SUMMARY:
Introduction: Parkinson's disease (PD) is the association of tremor, rigidity, akinesia-bradykinesia and loss of postural reflexes. Non-motor symptoms such as cognitive impairment may also develop. Cognitive impairment can be highly variable in its progression, symptoms and severity and can begin from the onset of the disease to the most advanced stages. Frailty is a syndrome characterized by a decrease in physiological reserve that results in an individual's increased vulnerability, which can lead to a variety of adverse factors when exposed to stressors. PD and frailty are highly prevalent in older people and are associated with increased morbidity and mortality. The presence of frailty in patients with PD is poorly studied, as is the association between cognitive impairment and frailty in this patient profile.

Objective: Evaluate the relationship between frailty and cognitive impairment in patients with PD or secondary parkinsonism.

Study design: observational, descriptive, correlative and cross-sectional.

Study population: The subjects that will be part of this study will be men and women with a diagnosis of PD or secondary parkinsonism belonging to the Health Area V of the Health Service of the Principality of Asturias, Spain.

DETAILED DESCRIPTION:
Introduction: Parkinson's disease (PD) is the association of tremor, rigidity, akinesia-bradykinesia and loss of postural reflexes. Non-motor symptoms such as cognitive impairment may also develop. Cognitive impairment in PD can be very varied in its progression, symptoms and severity, and can begin from the onset of the disease to the most advanced stages. At the same time, it may be one of the most prevalent non-motor symptoms in PD, with mild cognitive impairment being present in 20% to 30% of patients. Frailty is a syndrome characterized by a decrease in physiological reserve that results in an individual's increased vulnerability, which can lead to a variety of adverse factors when exposed to stressors. There are three prominent theoretical frameworks for the study of frailty, the physical model developed by Fried et al., the deficit accumulation model by Rockwood et al. and the biopsychosocial model by Gobbens et al. PD and frailty are highly prevalent in older people and are associated with increased morbidity and mortality. The presence of frailty in patients with PD is poorly studied, as is the association between cognitive impairment and frailty in this patient profile.

Objective: Evaluate the relationship between frailty and cognitive impairment in patients with PD or secondary parkinsonism.

Study design: observational, descriptive, correlational and cross-sectional.

Study population: The subjects that will be part of this study will be men and women with a diagnosis of PD or secondary parkinsonism belonging to the Health Area V of the Health Service of the Principality of Asturias, Spain.

Data collection: Data will be collected by means of a structured, face-to-face interview at the patient's home or at the Jovellanos Parkinson's Association facilities. These assessments will be carried out, whenever possible, in the presence of a family member or the patient's primary caregiver. The collection of information, the assessment of the patients and the completion of the questionnaires will be carried out by two physiotherapists who are experts in home care following the same guidelines and applying exactly the same criteria.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, without age limit, with a diagnosis of PD or secondary parkinsonism.
* Patients belonging to Health Area V of the Health Service of the Principality of Asturias, Spain.
* Patients who have been referred to the Home Rehabilitation Service of the Instituto de Rehabilitación Astur S.A. and/or who belong to the Jovellanos de Gijón Parkinson's Association of Gijón.
* Obtaining a score of more than 24 points in the Mini Mental State Examination (MMSE).
* Signing the informed consent form.

Exclusion Criteria:

* Parkinsonisms plus or atypical (progressive supranuclear palsy, multiple system atrophy, corticobasal degeneration, Lewy body disease).
* Acute disease causing clinical instability.
* Stage 5 of the Hoehn and Yahr scale.
* Patients unable to speak.
* Terminally ill patients.
* Patient with dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men and women diagnosed with PD or secondary parkinsonism
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Frailty: Fried's Frailty Phenotype | Baseline
  Fried's Frailty Phenotype proposed in the Cardiovascular Health Study consists of 5 criteria: unintentional weight loss, exhaustion, low physical activity, reduced grip strength, and reduced gait speed. It has a total score ranging from 0 to 5. A frail person is who scores 3 to 5; prefrail when scores 1 to 2, and robust when scores 0.
Frailty: Clinical Frailty Scale. | Baseline
  The Clinical Frailty Scale (CFS) was proposed in the Canadian Study of Health and Aging. It is a hierarchical scale of 9 levels ranging from 1, the best state of health, to 9, the worst situation: fit, well, well managed, vulnerable, mildly frail, moderately frail, severely frail, very severely frail, terminally ill.
Cognitive function: Parkinson's Disease Cognitive Rating Scale (PD-CRS). | Baseline
  Parkinson's Disease Cognitive Rating Scale (PD-CRS): It is a scale designed to detect the entire spectrum of cognitive dysfunction that occurs in the course of PD. It consists of nine cognitive tasks distributed in two sub-scores, with a maximum score of 134 points: fronto-subcortical (fixation verbal memory 12 points, maintained attention 10 points, working memory 10 points, drawing a clock 10 points, deferred verbal memory 12 points, alternating verbal fluence 20 points, action verbal fluence 30 points) and posterior cortical (denomination by confrontation 20 points and copy of a clock 10 points).

SECONDARY OUTCOMES:
Education level | Baseline
  Maximum level of education attained. Qualitative variable in 5 categories: illiterate (cannot read or write), no education (incomplete primary education), complete primary education, secondary education and university education.
Duration of the disease | Baseline
  The number of months since the patient was diagnosed with Parkinson's disease or Parkinsonism will be recorded.
Polypharmacy | Baseline
  Number of different drugs normally taken by the patient assessed in 24 hours. The consumption of more than 6 drugs will be considered polymedication.
Number of falls | Baseline
  The number of falls suffered in the last year will be collected.
Comorbidities | Baseline
  It is evaluated according to the Charlson comorbidity index. This scale consists of 19 items. Absence of comorbidity between 0 and 1 points, low comorbidity 2 points, high comorbidity between 3 and 5 points and severe comorbidity more than 5 points is considered.
Hoehn and Yahr scale | Cross-sectional baseline
  This scale indicates the degree of severity of the disease. It is divided into 6 states. Part of State 0 where there are no symptoms of the disease, until State 5 where the patient is totally dependent.
Movement Disorder Society Unified Parkinson´s Disease Rating Scale (MDS-UPDRS). | Baseline
  This tool allows to study the symptoms and the evolution of the disease. It is a scale that is subdivided into 4 parts. Part I: non-motor experiences of daily life, comprising 13 items; Part II: motor experiences of daily life, comprising 13 items; Part III: motor exploration, covering 18 items; and Part IV: motor complications, including 6 items. Each question is evaluated from 0 to 4, where 0 is normal and 4 the greater severity, the higher the score the greater involvement (greater impact of PD symptoms).
Quality of life. PDQ-39 | Baseline
  The Spanish version of the questionnaire Parkinson s disease quality of life questionnaire (PDQ39) is used. It consists of 39 items with 5 possible answers. 8 dimensions are analyzed: mobility, daily life activities, emotional well-being, stigma, social support, cognitive impairment, communication and body discomfort. The higher the score, the greater the impact on quality of life.
Barthel Index | Baseline
  Functional independence is measured using the Barthel index. It has a total score ranging from 0 to 100, where 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
Lawton Brody Index | Baseline
  Functional independence is measured with the Lawton and Brody Questionnaire. Instrumental activities of daily living assesses the ability to use the telephone, shop, use transport, cook, do household chores, take medication and manage finances. It has a total score ranging from 0 to 8, with 0 indicating total dependence and the maximum score indicating total independence.
SPPB activity level | Baseline
  Physical performance is measured using the Brief Physical Performance Battery. This measure consists of walking 4 m, a balance test with 3 levels (tandem, semi-tandem and feet together) and sitting and reaching 5 times as fast as possible. Total scores range from 0 to 12, with higher scores denoting higher physical performance.
Timed Up and Go (TUG) | Baseline
  Assesses balance, walking difficulties and decreased strength in lower limbs. This test consists of asking the person to get up from a chair with armrests, walk 3 meters, back and sit again, timing the time spent. 10 seconds or less: correct time. Between 10 and 20 seconds: frail marker. Between 20 and 30 seconds risk of falling. More than 30 seconds: high risk of falls.
Walking evaluation FAC | Baseline
  It is measured according to the Holden Ambulation Classification (FAC). It consists of 6 response categories, from the value 0 (no gear) to the value 5 (independent gear including up and down stairs).

CONTACTS AND LOCATIONS:
Overall Officials: MC Sousa-Fraguas, Principal Investigator — University of Oviedo
Locations (1):
- Home patients, Gijón, Principality of Asturias, Spain

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Background] Gobbens RJ, van Assen MA, Luijkx KG, Wijnen-Sponselee MT, Schols JM. The Tilburg Frailty Indicator: psychometric properties. J Am Med Dir Assoc. 2010 Jun;11(5):344-55. doi: 10.1016/j.jamda.2009.11.003. Epub 2010 May 8. PMID 20511102
- [Background] Pagonabarraga J, Kulisevsky J, Llebaria G, Garcia-Sanchez C, Pascual-Sedano B, Gironell A. Parkinson's disease-cognitive rating scale: a new cognitive scale specific for Parkinson's disease. Mov Disord. 2008 May 15;23(7):998-1005. doi: 10.1002/mds.22007. PMID 18381647
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Granger CV, Albrecht GL, Hamilton BB. Outcome of comprehensive medical rehabilitation: measurement by PULSES profile and the Barthel Index. Arch Phys Med Rehabil. 1979 Apr;60(4):145-54. PMID 157729
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Holden MK, Gill KM, Magliozzi MR, Nathan J, Piehl-Baker L. Clinical gait assessment in the neurologically impaired. Reliability and meaningfulness. Phys Ther. 1984 Jan;64(1):35-40. doi: 10.1093/ptj/64.1.35. PMID 6691052
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Derived] Sousa-Fraguas MC, Rodriguez-Fuentes G, Lastra-Barreira D, Conejo NM. Associations between frailty and cognitive impairment in Parkinson s disease: a cross-sectional study. Aging Clin Exp Res. 2025 Jan 3;37(1):19. doi: 10.1007/s40520-024-02922-4. PMID 39751989